CLINICAL TRIAL: NCT05019820
Title: Identification of Sarcopenia in Knee Osteoarthritis With Ultrasonography and Evaluation of Muscle Architecture Change by Ultrasonography After Isokinetic Exercise Program
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sema Dağcı (Other)
Responsible Party: Sponsor-Investigator, Sema Dağcı, Principal Investigator, Mustafa Kemal University
Organization: Mustafa Kemal University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MustafaKU-Sar-KOA
Record Dates: First submitted 2021-07-23; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Osteoarthritis of the Knee; Sarcopenia
MeSH Terms: conditions — Osteoarthritis, Knee; Sarcopenia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sarcopenia and osteoarthritis group (Active Comparator): Women aged 45-65 years diagnosed with sarcopenia and knee osteoarthritis
  Interventions: Other: Knee strengthening exercises with isokinetic dynamometer
- Without osteoarthritis and sarcopenia group (Other): Women aged 45-65 years without a diagnosis of knee osteoarthritis and sarcopenia
  Interventions: Other: Strengthening around the knees with home exercise programe

INTERVENTIONS:
Other: Knee strengthening exercises with isokinetic dynamometer — 18 sessions of strengthening exercises around the knee with an isokinetic dynamometer 3 days a week
  Arms: Sarcopenia and osteoarthritis group
Other: Strengthening around the knees with home exercise programe — 18 sessions of strengthening exercises for the muscles around the knee at home, 3 days a week
  Arms: Without osteoarthritis and sarcopenia group

SUMMARY:
The aim of this thesis; To define sarcopenia in knee osteoarthritis with ultrasonography and to evaluate changes in muscle structure in sarcopenia after isokinetic exercise application ultrasonographically. The investigators will evaluate the effect of isokinetic exercise therapy in sarcopenic patients with knee osteoarthritis with VAS (Visual Analog Scale) and WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index). Then, the hand grip strength will be evaluated with a dynamometer, and its effects on physical performance will be evaluated by 6 meters walking and chair rising tests.

DETAILED DESCRIPTION:
Among the 45-65 age group who applied to Mustafa Kemal University Faculty of Medicine, Physical Medicine and Rehabilitation outpatient clinic, 30 female patients diagnosed with knee osteoarthritis (stage 1-2-3) and sarcopenia together, and 30 individuals without osteoarthritis and sarcopenia will be included in the study as the control group.Patients with knee osteoarthritis who have been diagnosed with sarcopenia by ultrasonography will be Group I, and the control group without osteoarthritis and sarcopenia will be Group II.30 patients in Group I will be given an exercise program with isokinetic dynamometer for both knees, 30 minutes of TENS (transcutaneous electrical nerve stimulation), 20 minutes of hot packs, and home exercise program will be given lower extremity strengthening for a total of 6 weeks (18 sessions), 3 sessions per week.A diet program (protein, mineral, vitamin D supplemented) will also be given to these patients. The control group, which is group II, will be offered a home exercise program and diet for lower extremity strengthening only.Those with a history of complicated Diabetes Mellitus, Severe Coronary Artery Disease / Congestive Heart Failure, severe Liver Failure, neuromuscular disease, previous lower extremity surgery, rheumatological disease, use of walking aids will not be included in the study.The patient group and control group pre-treatment (week 0) and post-treatment (week 6) clinical; hand grip strength will be evaluated with Jamar dynamometer, walking speed will be evaluated with 6 meters walking test, lower extremity endurance will be evaluated with chair rise test, functional assessment of knee osteoarthritis will be evaluated by WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) and pain assessment will be evaluated by VAS (Visual Analogue scale) will be evaluated with a pain questionnaire.In addition, changes in the Rectus Femoris and Vastus Lateralis muscle architecture on the dominant side of the patients; muscle thickness, fascicle length, echogenicity, pennation angle and cross-sectional area measurements will be evaluated before treatment (0 weeks) and after treatment (6 weeks) by ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Among the 45-65 age group, 30 female patients diagnosed with knee osteoarthritis (Stage 1-2-3) and sarcopenia together
* Among the 45-65 age group, 30 females without osteoarthritis and sarcopenia will be included in the study as the control group.

Exclusion Criteria:

* Diabetes Mellitus,
* Severe Coronary Artery Disease / Congestive Heart Failure,
* Severe Liver Failure,
* Neuromuscular disease,
* Lower extremity surgery,
* Rheumatological disease,
* Those who use walking aids

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2021-11-20 (Estimated); Study Completion 2022-12-13 (Estimated)

PRIMARY OUTCOMES:
Muscle architecture | Six weeks
  Determination of muscle architecture change with ultrasonography after isokinetic exercise

SECONDARY OUTCOMES:
Knee pain | Six weeks
  The effect of isokinetic exercise with VAS (visual analog scale) on pain level
Functional status | Six weeks
  Effect of isokinetic exercise on activities of daily living with WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index)
Hand grip strength | Six weeks
  Evaluating the effect of isokinetic exercise on hand grip strength with a hand dynamometer
Walking speed | Six weeks
  Evaluation of the change in walking speed with isokinetic exercise
Time to get out of the chair | Six weeks
  Evaluation of the change in sitting time by standing up from the chair 5 times with isokinetic exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal University, Hatay, Antakya, Turkey (Türkiye)

REFERENCES:
- [Background] Spinoso DH, Bellei NC, Marques NR, Navega MT. Quadriceps muscle weakness influences the gait pattern in women with knee osteoarthritis. Adv Rheumatol. 2018 Aug 31;58(1):26. doi: 10.1186/s42358-018-0027-7. PMID 30657091
- [Background] Lange AK, Vanwanseele B, Fiatarone Singh MA. Strength training for treatment of osteoarthritis of the knee: a systematic review. Arthritis Rheum. 2008 Oct 15;59(10):1488-94. doi: 10.1002/art.24118. PMID 18821647
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Kara M, Kaymak B, Ata AM, Ozkal O, Kara O, Baki A, Sengul Aycicek G, Topuz S, Karahan S, Soylu AR, Cakir B, Halil M, Ozcakar L. STAR-Sonographic Thigh Adjustment Ratio: A Golden Formula for the Diagnosis of Sarcopenia. Am J Phys Med Rehabil. 2020 Oct;99(10):902-908. doi: 10.1097/PHM.0000000000001439. PMID 32941253
- [Background] Papalia R, Zampogna B, Torre G, Lanotte A, Vasta S, Albo E, Tecame A, Denaro V. Sarcopenia and its relationship with osteoarthritis: risk factor or direct consequence? Musculoskelet Surg. 2014 Jun;98(1):9-14. doi: 10.1007/s12306-014-0311-6. Epub 2014 Jan 31. PMID 24482109
- [Background] Baroni BM, Geremia JM, Rodrigues R, De Azevedo Franke R, Karamanidis K, Vaz MA. Muscle architecture adaptations to knee extensor eccentric training: rectus femoris vs. vastus lateralis. Muscle Nerve. 2013 Oct;48(4):498-506. doi: 10.1002/mus.23785. Epub 2013 Jul 15. PMID 23852989
- [Result] Lespasio MJ, Piuzzi NS, Husni ME, Muschler GF, Guarino A, Mont MA. Knee Osteoarthritis: A Primer. Perm J. 2017;21:16-183. doi: 10.7812/TPP/16-183. PMID 29035179